CLINICAL TRIAL: NCT01549639
Title: Use of a Novel Point of Care Device to Measure Blood Propofol Levels During Propofol Based General Anesthesia by Target Controlled Infusion Using the Marsh Model in Effect Site Mode
Brief Title: Blood Propofol Measurement During Anaesthesia Using Propofol Target Controlled Infusion
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nicholas J Cowley, Lead investigator, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: rrk4342
Record Dates: First submitted 2012-03-02; First posted 2012-03-09 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: General Anaesthesia; Propofol; Target Controlled Infusion; Pharmacokinetics
Keywords: Propofol; Target controlled infusion; General anaesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- General Anaesthesia: Patients undergoing general anaesthesia using Marsh model target controlled infusion in effect site mode.

SUMMARY:
Propofol is a commonly used agent for sedation and anaesthesia in the intensive care unit and the operating room. The pharmacokinetics of propofol are difficult to predict in patients not conforming to the norms in which the original pharmacokinetic research was based. Such patients, including the critically ill, and morbidly obese, are increasingly being encountered. The investigators group have been involved in the development of a device which can measure blood propofol concentrations, and hope for this to be available to use in the operating room in a clinically useful timeframe in the future. Data will be collected on patients undergoing propofol based general anaesthesia. The Marsh target controlled algorithm in effect site mode (commonly used by anaesthetists) will be assessed for accuracy using the propofol monitor. A new proportional correction method will be developed using this data, designed to enable recalibration of the TCI algorithm in near real time in order to achieve a more accurate estimated propofol concentration in these identified patient groups. The research will investigate the effectiveness of a correction of estimated propofol levels based on a one off measurement early on in the anaesthetic, and will take subsequent samples to measure propofol levels without modifying the TCI algorithm. Additionally, data on anaesthetist choice of TCI model, and method of administration in this relatively unselected group of patients will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Only patients undergoing major surgery where blood sampling through arterial or central venous catheters is part of their routine clinical care will be recruited.
* Only patients undergoing total intravenous anaesthesia using propofol will be recruited.

Exclusion Criteria:

* Anaemic patients will not be recruited into the study.
* Patients unable to consent will not be recruited into the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in the Operating Theatre undergoing propofol intravenous anaesthesia who require an arterial line to be inserted as standard care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Median percentage prediction error of estimated propofol concentration compared to measured concentrations (Bias) | duration of anaesthesia (up to 24 hours)

SECONDARY OUTCOMES:
Median absolute percentage prediction error of estimated propofol concentration compared to measured concentrations (inaccuracy) | duration of anaesthesia (up to 24 hours)
Change in median percentage prediction error(bias)for propofol levels measured beyond thirty minutes following proportional correction at thirty minutes | thirty minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Cowley, MRCP FRCA, Principal Investigator — University Hospital Birmingham NHS Foundation Trust; Thomas Clutton-Brock, FRCA FRCP, Study Chair — University Hospital Birmingham NHS Foundation Trust
Locations (1):
- University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands, United Kingdom